CLINICAL TRIAL: NCT00087412
Title: Phase II Trial of OSI-774 (NSC-718781) in Patients With Advanced Non-Small Cell Lung Cancer and a Performance Status of 2
Brief Title: S0341: Erlotinib in Treating Patients With Advanced Primary Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03060; S0341; U10CA032102 (NIH); CDR0000377245 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Adenocarcinoma of the Lung; Large Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (1):
- Treatment (Experimental): Patients receive oral erlotinib once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well erlotinib works in treating patients with advanced primary non-small cell lung cancer. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess survival in patients with advanced non-small cell lung carcinoma with a Zubrod Performance Status of 2 treated with OSI-774.

II. To evaluate the objective tumor response rates (confirmed plus unconfirmed, complete and partial), in patients with advanced non-small cell lung carcinoma with a Zubrod Performance Status of 2 treated with OSI-774.

III. To investigate in a preliminary manner possible correlations of EGFR expression, mutations, and/or EGFR polymorphisms with response and/or survival.

IV. To investigate in a preliminary manner possible correlations of activated signal pathway molecules, including basal p27 expression levels with response and/or survival.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven newly diagnosed selected stage IIIB (T4 lesion due to malignant pleural effusion) or stage IV, advanced primary non-small cell lung cancer (adenocarcinoma, large cell carcinoma, squamous cell carcinoma or unspecified) or recurrent disease after previous surgery and/or irradiation
* Patients with brain metastases are ineligible; all patients with neurological abnormalities on physical exam or symptoms must have a negative pretreatment CT or MRI scan of the brain within 28 days prior to registration
* Patients must have measurable disease documented by CT, MRI, X-ray, physical exam or nuclear exam within 28 days prior to registration; non-measurable disease must be assessed within 42 days prior to registration
* Patients must have a Zubrod performance status of 2
* Patients may have received prior radiation therapy provided that at least three weeks have elapsed since the completion of prior radiation therapy and patients have recovered from all associated toxicities; measurable disease must be present outside the previous radiation field or a new lesion must be present
* Patients may have received prior surgery provided that at least three weeks have elapsed since surgery (thoracic or other major surgeries) and patients have recovered from all associated toxicities; patients must have measurable residual disease present outside the area of surgical resection
* Patients must not have received prior hormonal, systemic (chemotherapy) or biologic therapy for non-small cell lung cancer; patients must not have received prior therapy with EGFR inhibitors
* Patients must not be currently receiving or planning to receive concurrent hormonal, biologic or radiation therapy to measurable or non-measurable lesions except patients may receive concurrent palliative radiation therapy to small field non-measurable sites of disease (painful bony metastases) as long as there are other sites of measurable disease outside of the radiation treatment field
* ANC of >= 1,500/ul
* Platelet count of >= 100,000/ul
* Serum bilirubin =< the institutional upper limit of normal (IULN) AND must satisfy one of the following:

  * Alkaline phosphatase =< IULN and liver enzymes (SGOT or SGPT) =< 2 x the IULN
  * Alkaline phosphatase =< 4 x the IULN and liver enzymes (SGOT or SGPT) =< the IULN
* Serum creatinine =< 2 mg/dl
* Patients must not have gastrointestinal tract disease resulting in an inability to take enteral medication, malabsorption syndrome, a requirement for IV alimentation, had prior surgical procedures affecting absorption or uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Patients must have completed the prestudy Medical Conditions Questionnaire

  * Patients are not required to complete the Medical Conditions Questionnaire if they are unable to read and understand English
* Correlative science studies: institutions must have received IRB approval of S9925 (the Lung Cancer Specimen Repository); patients must be offered participation in S9925; with the patient's consent, blood, plasma and tissue will be submitted for testing via S9925; patients must be registered separately to S9925 in order for institutions to receive credit for specimen submission
* Patients must not have a significant history of cardiac disease, i.e., uncontrolled high blood pressure, unstable angina, congestive-heart failure, myocardial infraction within the last six months, or cardiac ventricular arrhythmias requiring medication
* Patients must be willing to provide prior smoking history
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* If day 14, 28 or 42 falls on a weekend or holiday, the limit may be extended to the next working day

  * In calculating days of tests and measurements, the day a test or measurement is done is considered day 0; therefore, if a test is done on a Monday, the Monday four weeks later would be considered day 28; this allows for efficient patient scheduling without exceeding the guidelines
* Pregnant or nursing women may not participate in this trial; women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-09; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Median survival | Up to 3 years

SECONDARY OUTCOMES:
Response rates (confirmed plus unconfirmed, complete plus partial) | Up to 3 years
Toxicity rates graded according to the NCI CTCAE version 3.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hesketh, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States